CLINICAL TRIAL: NCT04733872
Title: Using Vegetable and Berry Products Can Improve Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180905VAB
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases | interventions — Vegetables

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): subjects drank 50 ml , 1 bottle a day for 8 week
  Interventions: Dietary Supplement: placebo
- Vegetable and Berry Drink (Experimental): subjects drank 50 ml , 1 bottle a day for 8 week
  Interventions: Dietary Supplement: Vegetable and Berry Drink

INTERVENTIONS:
Dietary Supplement: placebo — subjects drank 50 ml , 1 bottle a day for 8 week
  Arms: placebo group
Dietary Supplement: Vegetable and Berry Drink — subjects drank 50 ml , 1 bottle a day for 8 week
  Arms: Vegetable and Berry Drink

SUMMARY:
Hypothesis: vegetable and berry products for 8 weeks can improve skin condition

DETAILED DESCRIPTION:
Hypothesis: Using vegetable and berry products for 8 weeks can improve skin condition

ELIGIBILITY:
Inclusion Criteria:

1. Dry skin
2. Rough skin
3. Large pores
4. Dark yellow complexion
5. Sagging skin

Exclusion Criteria:

1. Skin disorders
2. Liver diseases
3. Kidney diseases
4. Allergy to cosmetics, drugs, or foods
5. Pregnant and lactating women
6. People who had any cosmetic procedures before 4 weeks of the study
7. Area of facial spot over 3 cm2
8. Vegan
9. People who took collagen supplements in the past 3 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
skin moisture | up to 8 week
  using corneometer CM825 to examine skin moisture (The higher the value, the more water content, C.U., corneometer units ).subjects drank 50 ml after meal
skin elasticity | up to 8 week
  using cutometer dual MPA580 to examine skin elasticity (The closer the R2 value is to 1, the better the elasticity and no unit)
skin gloss | up to 8 week
  using probe system GL2000 & MPA10 to examine skin gloss (The higher the value, the higher the gloss, no unit)
skin spot | up to 8 week
  usig VISIA-CR to examine skin spot (The higher the value, the larger the pore area, mm2)
skin wrinkle | up to 8 week
  using VISIOSCAN-VC20 to examine skin wrinkle (The higher the value, the more wrinkles, surface evaluation of wrinkles, SEW)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Research & Design Center, TCI CO., Ltd, Taipei, Neipu Township, Taiwan

IPD SHARING:
Plan to Share IPD: No